CLINICAL TRIAL: NCT04108494
Title: A Single-center, Randomized, Controlled Trial to Evaluate Total Versus Partial Omentectomy for Advanced Gastric Cancer in Radical Gastrectomy
Brief Title: A Trial of Total Versus Partial Omentectomy for Advanced Gastric Cancer in Gastrectomy
Acronym: TOP1
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E2019054
Record Dates: First submitted 2019-09-15; First posted 2019-09-30 (Actual); Last update posted 2019-09-30 (Actual); Status verified 2019-09

CONDITIONS: Gastric Cancer
Keywords: Gastric Cancer; Omentectomy; Prognosis
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): D2 radical gastrectomy with partial omentectomy
  Interventions: Procedure: Type of omentectomy
- Control group (No Intervention): D2 radical gastrectomy with total omentectom

INTERVENTIONS:
Procedure: Type of omentectomy — Partial omentectomy with preservation of the greater omentum at >3 cm from the gastroepiploic arcade.Control group with total omentectomy.
  Arms: Experimental group

SUMMARY:
The main purpose of this study is to evaluate the impact of omentectomy for advanced gastric cancer on patient survival.

DETAILED DESCRIPTION:
Surgical resection is the mainstay of treatment for gastric cancer. The extent of surgical resection includes total or subtotal gastrectomy, D2 lymphadenectomy, and prophylactic or therapeutic resection of the surrounding organs or tissues (e.g., omentum, peritoneum, etc). However, the oncologic importance of omentectomy during gastrectomy remains unclear. The European guidelines do not give any advice regarding omentectomy, whereas the most recent American guidelines advise to resect both the greater and lesser omentum. Alternatively, the Japanese gastric cancer treatment guidelines recommends preservation of the greater omentum at >3 cm from the gastroepiploic arcade for patients with T1-T2 tumors and total omentectomy for patients with T3-T4 tumors. In order to evaluate the impact of omentectomy for advanced gastric cancer on patient survival, we designed this trial. Patients who received curative gastrectomy were divided into two groups based on whether they underwent omentectomy. The primary endpoint is the 3-year relapse-free survival rate and the secondary endpoints are 5-year overall survival, and postoperative morbidity.

ELIGIBILITY:
Inclusion Criteria:

1. Had been treated with Radical resection (D2, R0) of gastric cancer (Lymph node≥16);
2. Physical condition and organ function allows to tolerable abdominal surgery;
3. Willing and able to comply with the program during the study period;
4. Written informed consent provided;
5. ≥ 18 and ≤ 70 years of age; preoperative gastric cancer patients with pathologically confirmed;
6. With more than a 6-month life expectancy;
7. No other serious concomitant diseases; Sufficient organ functions;
8. No previous history of chemotherapy or radiotherapy;
9. All patients accept 8 cycles XELOX chemotherapy regimen;
10. Clinical stage: T2-4aN0-+M0;
11. Macroscopic types :Borrmann I-III;
12. Not greater curvature tumor;
13. No previous surgery for any abdominal disease, except an appendectomy for appendicitis, a laparoscopic cholecystectomy for gallbladder stones; No previous history of peritonitis, pancreatitis;
14. Karnofsky performance status (KPS)>60; Eastern Cooperative Oncology Group Performance Status (ECOG): 0-1.

Exclusion Criteria:

1. Pregnancy or breast feeding;
2. Patients with Serious liver disease (such as cirrhosis, etc.), kidney disease, respiratory disease or uncontrolled diabetes, hypertension and other chronic systemic diseases, heart disease with Clinical symptoms, such as congestive heart failure, coronary heart disease symptoms, drug is difficult to control arrhythmia, hypertension, or six months had a myocardial infarction attack, or cardiac insufficiency;
3. Organ transplantation patients need immunosuppressive therapy;
4. Severe recurrent infections were not controlled or with other serious concomitant diseases;
5. Patients got other primary malignant tumors (except curable skin basal cell carcinoma and cervical cancer in situ) except gastric cancer within 5 years;
6. Psychiatric disease which require treatment;
7. Have the history of organ transplantation;
8. Within 6 months before study starts and in the process of this study, patients participate in other clinical researches.
9. Advanced gastric cancer with omentum invasion
10. Patients can't treated with XELOX after surgery;
11. Macroscopic types : Borrmann IV;
12. Tumor invasion of adjacent organ (T4b) or with distant metastasis（M1）;
13. Tumor invasion the greater curvature invasion.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 418 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
3 years relapse-free survival | 3 years
  Relapse-free survival l (RFS) was defined as the length of time from the date of randomization to the date of first documentation of relapse of gastric cancer or any other type of cancer or death.

SECONDARY OUTCOMES:
5 years overall survival | 5 years
  Overall survival (OS) was defined as the length of time from the date of randomization to the date of death of various reasons.

OTHER OUTCOMES:
The volume of intraoperative blood loss | 1 week
  The volume of intraoperative blood loss (IBL) was defined as the total from suction and the weight of gauze sponges at the conclusion of the operation. The Blood loss volume is recorded in milliliters.
The length of the operation | 1 week
  The length of the operation was defined as the time from first skin incision to wound closure. The length of the operation is recorded in minutes.
Postoperative hospital stay | 3 months
  Postoperative hospital stay was defined as the time from the date of operation to the date of discharge. The postoperative hospital stay is recorded in days.
Postoperative morbidity | 1 month
  Postoperative morbidity was defined as the incidence rate of the postoperative complication. The postoperative morbidity were examined within 30 days after surgery. Postoperative morbidity was graded with use of the modified Clavien-Dindo classification of surgical complications.

CONTACTS AND LOCATIONS:
Overall Officials: Han Liang, Master, Study Chair — Tianjin Medical University Cancer Institute and Hospital
Locations (1):
- Tianjin Medical University Cancer Hospital, Tianjin, Tianjin Municipality, China